CLINICAL TRIAL: NCT02934893
Title: A Randomized, Controlled, Open-label, Multi-center Study to Evaluate the Effect and Benefit of Diabetes Management Decision Support Software for Blood Glucose Control
Brief Title: A Study to Evaluate the Effect and Benefit of Diabetes Management Decision Support Software for Blood Glucose Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rimidi Diabetes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RD-DOHC
Record Dates: First submitted 2016-08-17; First posted 2016-10-17 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intervention Group (Experimental): Patient in standard diabetes management in the Medication Management Clinic plus the use of Diabetes+Me plus connected glucometer
  Interventions: Other: Medication Management Clinic; Other: Diabetes+Me plus connected glucometer
- Standard Diabetes Management (Active Comparator): Patient in standard diabetes management in the Medication Management Clinic
  Interventions: Other: Medication Management Clinic
- Primary Care (No Intervention): Matched cohort managed through their primary care physician (PCP) and standard of care.

INTERVENTIONS:
Other: Medication Management Clinic — referral to medication management clinic from primary care
  Arms: Intervention Group; Standard Diabetes Management
Other: Diabetes+Me plus connected glucometer — Use of software and medication modeling tool as add on to medication management standard of care
  Arms: Intervention Group

SUMMARY:
The benefit of drug therapy to persons with diabetes has been well established in clinical trials in terms of reducing cardiovascular risk, microvascular complications and mortality. However, treatment adherence and treatment effectiveness continue to be challenges in diabetes management.

Rimidi Diabetes has developed software algorithms to simulate the effect of anti-diabetic medications on an individual's glucose profile, allowing the clinician and their patient to visualize the anticipated outcome of a medical intervention. Use of this technology should allow for more targeted decision-making by the clinician and should facilitate a shared decision-making process with the PwD who is now privy to the thought process behind their medical management.

The proposed study is designed to test whether adding a decision support capability (Diabetes+Me Rx) that allows for modeling the anticipated effect of medication adjustments leads to improved glycemic control and a perceived benefit by healthcare providers and PwDs.

DETAILED DESCRIPTION:
* Recruitment

  * Recruitment of persons with diabetes through a community diabetes management center according to inclusion and exclusion criteria below.
  * This is a three-armed study. Enrollees will be randomized to continue diabetes care with standard diabetes management in the Medication Management Clinic or the Intervention Group and compared to a matched cohort managed through their primary care physician (PCP) and standard of care.
  * The Intervention Group will be standard diabetes management in the Medication Management Clinic plus the use of Diabetes+Me with a connected glucometer.
  * Upon recruitment, PwD will be oriented to the Diabetes+Me application and instructed on how to complete a glucose profile and how to enter data into the application. Baseline hemoglobin A1C will be measured.
  * Enrollees will complete a brief survey of satisfaction with their diabetes management.
* Study visits

  * The first study visit will be 2 weeks following enrollment.
  * Weight, number of medications, number of medication titrations, the presence of insulin and blood pressure will be measured at each study visit. Frequency of hypoglycemia in the preceding week will be documented at each visit. Adherence to medical prescription to be documented at each visit.
  * If the PwD has not entered data into Diabetes+Me this will be done at the beginning of each study visit.
  * At the first study visit, the HCP will review the glucose profile from the previous week, identify areas where the PwD is not meeting targets and model adjustments to their medications to achieve the desired anticipated effect. If indicated, a new prescription will be issued and the PwD instructed to collect a new glucose profile the week preceding the next visit.
  * The second study visit will occur 5 weeks following the initial visit. The HCP and PwD will review the glucose profile from the previous week, identify areas where the PwD is not meeting targets and model adjustments to their medications to achieve the desired anticipated effect. If indicated, a new prescription will be issued and the PwD instructed to collect a new glucose profile the week preceding the final visit.

The third and final study visit will occur 5 weeks following the second visit. The HCP and PwD will review the glucose profile from the previous week and identify if the PwD is meeting targets.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of type 1 or type 2 diabetes
* Glycated hemoglobin > 9% within 3 months
* Age 18-80
* Not currently managed by study clinicians

Exclusion Criteria:

* Pregnant
* Active substance abuse
* Severe hearing or visual impairment
* No internet or email access

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-10 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin A1C | change from baseline to 12 weeks

SECONDARY OUTCOMES:
Number of hypoglycemic events per week | change from 1st week to twelfth week
  Decrease in frequency of hypoglycemia (# events per week
Blood pressure | change from baseline to 12 weeks
  increase in percentage of patients with blood pressure in normotensive range
BMI | change from baseline to 12 weeks
  decrease in BMI
Healthcare provider satisfaction | through study completion, an average of 1 year
  healthcare provider satisfaction based on scoring of questionnaire
A1C target attainment | at 12 weeks
  time to A1c goal attainment
Medication titrations needed | 12 weeks
  number of medication titrations over 12 week period needed to reach A1c goal
Patient satisfaction questionnaire | through patient study completion, an average of 12 weeks
  questionnaire addresses satisfaction with care and knowledge of diabetes self-management

CONTACTS AND LOCATIONS:
Overall Officials: Michael Jardula, MD, Principal Investigator — Desert Oasis Healthcare

IPD SHARING:
Plan to Share IPD: Undecided